CLINICAL TRIAL: NCT07308665
Title: A Multi-site Retrospective Study of the Real-world Performance of Aquacel With Strengthening Fiber (WSF) Ribbon Dressings
Brief Title: Aquacel With Strengthening Fiber (WSF) Ribbon Dressings
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WC-24-450
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ulcer Foot; Ulcer Healing; Wound Infection
MeSH Terms: conditions — Foot Ulcer; Wound Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Aquacel Ribbon: Aquacel WSF Ribbon treatment
  Interventions: Device: Aquacel Ribbon

INTERVENTIONS:
Device: Aquacel Ribbon — Subjects who received an Aquacel WSF Ribbon

SUMMARY:
Retrospective, multi-site, non-comparative, post-market study

DETAILED DESCRIPTION:
Retrospective, multi-site, non-comparative, post-market study to evaluate real-world performance of Aquacel WSF Ribbon dressings in wound healing

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received one or more Aquacel WSF Ribbon dressing

Exclusion Criteria:

* Patients who have not received one or more Aquacel WSF Ribbon dressings

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received an Aquacel WSF Ribbon dressing and who's data was collected in Wound Care Advantage (WCA).
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Real-world efficacy of Aquacel WSF Ribbon in improving the incidence of wound closure | Baseline and week 4, 12, 20
  Time to complete wound closure, defined as 100% epithelialization of the wound surface

OTHER OUTCOMES:
Wound size | Baseline and week 4, 12, 20
  Measured size (area, volume) of target wound at each visit
Wound dept | Baseline and week 4, 12, 20
  Measured wound depth at each visit
Exudate volume | Baseline and week 4, 12, 20
  Changes in exudate volume
Application use | Up to week 20
  Number of Aquacel WSF Ribbon applications per subject over treatment course
Visit frequency | Up to week 20
  Number of visit frequency
Dressing wear time | Baseline and week 4, 12, 20
  Aquacel WSF Ribbon wear time

CONTACTS AND LOCATIONS:
Overall Officials: Christina Mastandrea, Study Director — ConvaTec Inc.